CLINICAL TRIAL: NCT04650828
Title: TDF Combined With LDT for the Treatment of HBeAg-positive Hepatitis B Patients With Poor Response to TDF for Twelve Months
Brief Title: TDF Combined With LDT for the Treatment of HBeAg-positive Hepatitis B Patients With Poor Response to TDF for 12 Months
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chaoshuang Lin, Professor Lin, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: 00000001
Record Dates: First submitted 2020-10-20; First posted 2020-12-03 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental:person with TDF+LDT: TDF combined with LDT for 12 months
  Interventions: Drug: TDF
- Active comparator:person with TDF: TDF monotherapy was continued for 12 months
  Interventions: Drug: Tenofovir Disoproxil Fumarate 300 MG

INTERVENTIONS:
Drug: TDF — TDF combined with telbivudine (LDT) for 12 months
  Groups: Experimental:person with TDF+LDT
Drug: Tenofovir Disoproxil Fumarate 300 MG — TDF monotherapy was continued for 12 months
  Groups: Active comparator:person with TDF

SUMMARY:
Studies have shown that the HBeAg seroconversion rate of HBeAg positive chronic hepatitis B with tenofovir for one year's treatment was 17.8% and the negative conversion rate of their HBeAg and HBV DNA were 20.0% and 97.6%. The HBeAg Seroconversion rate of these patients was lower.Clinically, most patients need to take tenofovir for a long time, which may cause serious complications such as renal function damage,with decreased therapy compliance and Increased cost of treatment.In the course of tenofovir treatment, it is common that HBV-DNA negative patients with HBeAg Being down poor or staying at a low positive level for a long time keep taking the medicine. Therefore, it is Significant to Increase the HBeAg seroconversion rate of tenofovir during the clinical treatment.

Telbivudine has a strong antiviral effect.Studies have shown that the HBeAg seroconversion rate of HBeAg positive CHB for one year was 25%, which was higher than other nucleosides, and it could also improve the damaged renal function to a certain extent.The HBeAg seroconversion rate of patients with poor response to tenofovir for 12 months could be still poor if for 24 months . Therefore, this study is to observe the efficacy of these patients combined with telbivudine.

DETAILED DESCRIPTION:
This is an open, multicenter, exploratory and real-world clinical study. It will be carried out in patients with poor response (HBV DNA > 2x103iu / ml) to tenofovir for 12 months. After one -week screening period, patients will be randomly assigned 1:1 to control and experimental groups. The control group takes tenofovir for 12 months while the experimental group takes tenofovir combined with telbivudinefor 12months .

ELIGIBILITY:
Inclusion criteria:

1. Male or female patients, aged 18 to 70 years, including 18 and 70 years old;
2. Patients with poor response to tenofovir for 12 months did not obtained HBeAg seroconversionPatients with poor response to tenofovir for 12 months who didn't obtain HBeAg seroconversion choosed to continue taking tenofovir or take tenofovir combined with Tbl for 12months;
3. Persons were willing to sign informed consent and comply with medication regimen and follow-up.

Exclusion Criteria:

1. Co-infectious with hepatitis A, hepatitis C, hepatitis D, hepatitis E or HIV;
2. In the decompensated stage of liver cirrhosis, such as ascites, varicose bleeding or hepatic encephalopathy;
3. With malignant tumors (including hepatocellular carcinoma);
4. Concomitant with other liver diseases, such as alcoholic liver disease, autoimmune disease, or other systemic diseases involving the liver, such as hemochromatosis, Alpha-1 antitrypsin deficiency, or Wilson disease;
5. During the study period, chronic systemic steroid drugs are required or may be used under any medical conditions;

There are any other factors that the researcher thinks are not suitable for inclusion in the study, or that may affect the patient's participation or completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with poor response (HBV DNA > 2x103iu / ml) to tenofovir for 12 months
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
HBeAg seroconversion rates | 12months
  HBeAg seroconversion rates at 12 months after tenofovir plus telbivudine treatment
HBeAg seroconversion rates | 24months
  HBeAg seroconversion rates at 24 months after tenofovir plus telbivudine treatment

SECONDARY OUTCOMES:
HBeAg negative rate | 12 and 24months
  HBeAg negative rate of tenofovir combined with telbivudine treatment at 12 and 24 months
ALT normalization rate | 12 and 24months
  ALT normalization rate of tenofovir combined with telbivudine treatment at 12 and 24 months
Renal function index | 12 and 24months
  Renal function index of tenofovir combined with telbivudine treatment at 12 and 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chaoshuang Lin, Guangzhou, China